CLINICAL TRIAL: NCT00562380
Title: A Phase 1, Open-Label, Dose Finding Study Evaluating the Safety and Pharmacokinetics of AMG 479 in Subjects With Advanced Solid Tumors
Brief Title: AMG-479 in Treating Patients With Advanced Solid Tumors or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AMGEN-479; CDR0000577404 (Registry Identifier: PDQ (Physician Data Query)); AMGEN-20050118; VU-VICC-050630; VU-VICC-PHI-0542
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2010-04

CONDITIONS: Lymphoma; Prostate Cancer; Sarcoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cutaneous B-cell non-Hodgkin lymphoma; angioimmunoblastic T-cell lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; small intestine lymphoma; splenic marginal zone lymphoma; unspecified adult solid tumor, protocol specific; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; adult desmoplastic small round cell tumor; recurrent adult soft tissue sarcoma; recurrent prostate cancer
MeSH Terms: conditions — Lymphoma; Prostatic Neoplasms; Sarcoma; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Neuroectodermal Tumors, Primitive, Peripheral; Desmoplastic Small Round Cell Tumor | interventions — ganitumab; Biopsy

INTERVENTIONS:
Biological: ganitumab
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as AMG-479, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of AMG-479 in treating patients with advanced solid tumors or non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and pharmacokinetics of anti-IGF-1R fully human monoclonal antibody AMG-479 (AMG-479) after multiple intravenous administrations in adult patients with histologically documented advanced solid tumors that are refractory to standard therapy or for which no curative therapy is available.

Secondary

* To assess the tolerability and to determine the maximum tolerated dose of AMG-479.
* To assess tumor glucose metabolism using PET/CT scanning with the tracer fludeoxyglucose F 18.
* To measure insulin-like growth factor receptor (IGF-1R) levels on peripheral blood cells.
* To establish whether human anti-human antibodies to AMG-479 develop in patients with advanced solid tumors.
* To measure the tumor response by modified Response Evaluation Criteria in Solid Tumors.

Tertiary

* To investigate bone turnover markers.
* To investigate potential biomarker development by biochemical analysis in blood cells and tumor cells.

OUTLINE: This is a multicenter study.

* Part 1 (dose-escalation): Patients receive escalating doses of anti-IGF-1R fully human monoclonal antibody AMG-479 (AMG-479) IV over 1 hour on days 1, 15, and 29. Patients are evaluated in week 8, and those who demonstrate an objective tumor response or stable disease continue treatment beginning on day 57. Treatment with AMG-479 repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
* Part 2 (randomized dose-expansion): Patients are randomized to one of two dose regimens.

  * Arm I: Patients receive AMG-479 IV over 1 hour at a lower dose on day 1.
  * Arm II: Patients receive AMG-479 IV over 1 hour at a higher dose on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity. Tumor tissue is obtained at baseline and after 4 weeks of study therapy for biomarker analysis.

Blood is drawn periodically for biomarker analysis (insulin-like growth factor [IGF]-1, IGF-binding protein 3 [IGF-BP3], IGF-1 receptor [IGF-1R], cross-linked c-telopeptides of type 1 collagen [CTx], bone-specific alkaline phosphatase [BSAP], and tartrate-resistant acid phosphatase [TRAP5b]) and pharmacokinetic studies.

After completion of study therapy, patients are followed for at least 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed advanced solid tumors or non-Hodgkin lymphoma that is refractory to standard treatment or for which no curative therapy is available
* Tumor tissue that is accessible for biopsy by using minimally invasive procedures and must consent to undergo biopsies of the tumor (part 2)

  * Exception for patients with Ewing family tumors or desmoplastic small round cell tumors whose anatomic location would pose an increase in the risk of injury due to biopsy (i.e., bleeding or pneumothorax)
* Willing to provide existing and/or future paraffin-embedded tumor samples

Exclusion criteria:

* Primary CNS tumors or hematological malignancies, other than non-Hodgkin lymphoma
* Primary hepatic tumors or at increased risk for hepatic tumors, including any of the following:

  * Hepatitis of any etiology
  * Alcohol abuse or dependency
  * Hepatic adenoma
  * Follicular nodular hyperplasia
  * Autoimmune conditions associated with biliary tract cancer
  * Alpha 1 antitrypsin deficiency
  * Hemochromatosis
  * History of vinyl chloride or thorotrast/thorium dioxide exposure
* History of histiocytic (Kupffer cell) neoplasia
* Presence of untreated or symptomatic CNS metastases or symptoms of brain metastases
* Presence of ascites or pleural effusion requiring medical intervention

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status ≤ 2
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to provide fasting blood samples for triglyceride and glucose laboratory tests
* Able to fast for 4-6 hours for fludeoxyglucose F18-PET/CT scan
* Controlled type 1 or 2 diabetes (defined as hemoglobin A1c < 8.0% and fasting blood glucose level < 160 mg/dL) allowed for part 2 only

Exclusion criteria:

* History of clinically significant hypoglycemia or hyperglycemia (in the opinion of the investigator)
* Myocardial infarction within the past year
* Unstable or uncontrolled disease/condition related to or impacting cardiac function, including any of the following:

  * Unstable angina
  * Congestive heart failure
  * NYHA class III or IV heart disease
  * Uncontrolled hypertension (diastolic BP > 90 mm Hg and systolic BP > 150 mm Hg)
  * Clinically significant cardiac arrhythmia
  * CTCAE version 3.0 ≥ grade 2
  * Clinically significant electrocardiogram abnormalities
* History of arterial or venous (deep vein) thrombosis within the past year
* History of bleeding diathesis
* History of chronic hepatitis
* History of HIV infection
* Unable to tolerate intravenous administration
* Known sensitivity to mammalian-derived products
* ANC < 1,500/mm^3 (without filgrastim [G-CSF] support within the past 2 weeks)
* Platelet count < 100,000/mm^3 (without transfusion within the past 2 weeks)
* Hemoglobin < 9 g/dL (without transfusion within the past 4 weeks)
* PT/PTT > 1.5 x upper limit of normal (ULN)
* Serum creatinine > 1.5 x ULN
* AST and ALT > 2.5 x ULN
* Total bilirubin > 1.5 x ULN
* Urinary protein excretion > 1,000 mg/day (≥ 2+ using dipstick analysis)
* Any kind of disorder that compromises the ability of the patient to give written informed consent and/or comply with study procedures
* Any comorbid medical condition, that in the sponsor's or investigator's opinion, may put the patients at significant risk
* Known sensitivity to any of the products to be administered during dosing
* Unresolved toxicities > grade 1 from prior anticancer therapy, excluding alopecia

PRIOR CONCURRENT THERAPY:

* No prior antitumor treatment within the past 28 days

  * Palliative external-beam radiotherapy to a lesion not used for RECIST measurement is acceptable during study for symptom management if patient is stable or improving and not progressing
* At least 30 days since prior and no concurrent enrollment in another clinical trial involving medication
* No antibody therapy for the treatment of underlying malignancy within the past 8 weeks
* No concurrent or prior anticoagulation therapy, except low-dose warfarin (< 2 mg/day) for prophylaxis against central venous catheter thrombosis
* No concurrent insulin (except diabetic patients enrolled in dose expansion [part 2] of the study)
* No other concurrent investigational procedures
* No concurrent blood or blood-product transfusions
* No concurrent herbal medications
* No other concurrent anticancer therapy including chemotherapy or hormonal therapy

  * Gonadotropic releasing-hormone agonists or antagonists allowed for advanced prostate cancer
* No major surgery within the past month and none planned for 28 days after completion of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2005-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety
Pharmacokinetic profile

SECONDARY OUTCOMES:
Level of insulin-like growth factor receptor-1 (IGF-1R) on peripheral blood cells
Tumor response measured by modified RECIST
Tumor glucose metabolism as measured by fludeoxyglucose F 18-PET/CT scan
Anti-AMG-479 antibody formation
The incidence of dose-limiting toxicities and the severity of adverse events
Levels of cross-linked c-telopeptides of type 1 collagen and bone-specific alkaline phosphatase (may also include tartrate-resistant acid phosphatase 5b) in blood
Circulating levels of IGF-1R and IGF-BP3

CONTACTS AND LOCATIONS:
Overall Officials: Mace L. Rothenberg, MD, FACP, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States